CLINICAL TRIAL: NCT06819566
Title: Prophylactic Endoscopic Variceal Ligation in Patients With High-risk Esophageal Varices Receiving Atezolizumab Plus Bevacizumab for Hepatocellular Carcinoma : A Phase II, Multicenter, Single-arm Trial (ESCOAT Trial)
Brief Title: Prophylactic Endoscopic Variceal Ligation in Patients With High-risk Esophageal Varices Receiving Atezo/Bev for HCC
Acronym: ESCOAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Hanyang University (Other); Samsung Medical Center (Other); National Cancer Center, Korea (Other Government); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ju Hyun Shim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1524
Record Dates: First submitted 2024-12-31; First posted 2025-02-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma; Esophageal Varix; Bleeding Esophageal Varices
Keywords: Hepatocellular carcinoma; Esophageal varix; Bleeding esophageal varices; Endoscopic variceal ligation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Esophageal and Gastric Varices

STUDY DESIGN:
Intervention Model Description: prophylactic EVL for high-risk esophageal varices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVL group (Experimental): This group is single arm which undergo prophylactic endoscopic variceal ligation for high-risk esophageal varices
  Interventions: Procedure: Endoscopic variceal ligation (EVL)

INTERVENTIONS:
Procedure: Endoscopic variceal ligation (EVL) — 1. EVL for high-risk varices will be performed by experienced endoscopists, certified in gastroenterological endoscopy, within two weeks prior to the initiation of the Atezo/Bev.
  2. A follow-up EGD will be conducted one week after the Atezo/Bev #3. If any of the following criteria are met, additional EVL will not be performed, and anticancer treatment will proceed two weeks later. Otherwise, an additional on-demand EVL session will be conducted:
     * The esophageal varices have improved to F1 or less.
     * The red color sign has disappeared.
  3. On-demand EVL will be considered after 5th, and 7th consecutive doses of Atezo/Bev, with EGD follow-up performed to assess eligibility. The maximum number of EVL sessions is limited to three sessions.

SUMMARY:
The goal of this study is to evaluate whether prophylactic endoscopic variceal ligation (EVL) can prevent esophageal variceal bleeding in patients with hepatocellular carcinoma (HCC) receiving atezolizumab and bevacizumab (Atezo/Bev) therapy. The study will also assess the safety of prophylactic EVL in this population.

The main question it aims to answer is:

Does prophylactic EVL in high-risk varices reduce the incidence of variceal bleeding to a level similar to that of low-risk varices in HCC patients receiving Atezo/Bev?

Participants will:

1. Undergo prophylactic EVL before starting Atezo/Bev therapy (within 2 weeks ± 1 week before the first dose).
2. Start Atezo/Bev therapy 2 weeks (± 1 week) after EVL.
3. Have follow-up endoscopies (EGD) one week after the 3rd, 5th, and 7th doses of Atezo/Bev.

If varices improve, no additional intervention is needed. If varices persist or worsen, on-demand EVL will be performed, and Atezo/Bev will continue.

This study will help determine if prophylactic EVL should be a standard strategy for managing high-risk varices in HCC patients undergoing Atezo/Bev therapy.

DETAILED DESCRIPTION:
1. Backgrounds Patients with hepatocellular carcinoma (HCC) undergoing treatment with atezolizumab plus bevacizumab (Atezo/Bev) are at a high risk of variceal bleeding. When bleeding occurs, it may necessitate treatment delays or permanent discontinuation of Atezo/Bev, potentially requiring a switch to alternative anticancer therapies that may be less effective. Additionally, variceal bleeding can result in hepatic decompensation, deteriorated liver function, and reduced quality of life.

   Prophylactic endoscopic variceal ligation (EVL) has been proposed as an approach to minimize the risk of variceal hemorrhage in patients with high-risk esophageal varices, as identified on screening endoscopy. By proactively treating high-risk varices before initiating Atezo/Bev, prophylactic EVL may optimize oncologic treatment continuity and overall patient outcomes.
2. Study aim

This Phase 2 study is designed to evaluate the efficacy and safety of prophylactic EVL in reducing variceal bleeding among HCC patients with high-risk esophageal varices undergoing Atezo/Bev therapy. In addition, this study aims to:

- Assess the impact of prophylactic EVL on patient survival and quality of life.

- Identify biomarkers associated with variceal bleeding risk and therapeutic response.

3. Study Design

1. Prophylactic EVL Procedure Prophylactic EVL will be performed within two weeks (± 1 week) before the initiation of Atezo/Bev therapy. The procedure will be conducted by board-certified gastroenterological endoscopists with expertise in therapeutic endoscopy.

   - EVL technique: Suctioning of esophageal varices until the red-out phenomenon occurs. Placement of a rubber band at the variceal base to induce thrombus formation, leading to subsequent necrosis and sloughing. The procedure begins at the distal esophageal varices and progresses spirally upward. Priority treatment will be given to varices with active bleeding or endoscopic signs of recent hemorrhage.
2. Follow-Up Endoscopy and Additional EVL Criteria Follow-up esophagogastroduodenoscopy (EGD) will be conducted one week after the 3rd dose of Atezo/Bev to assess variceal status.

   If any of the following criteria are met, additional EVL will not be performed, and Atezo/Bev therapy will continue two weeks later:
   * Varices have regressed to F1 or less
   * Red color signs have disappeared If these criteria are not met, an on-demand EVL session will be performed.
3. Further On-Demand EVL Strategy Additional on-demand EVL sessions will be considered after the 5th and 7th doses of Atezo/Bev, with EGD follow-up before each session.

The maximum number of EVL sessions will be limited to three during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older and under 80 years.
* Patients with liver function are classified as Child-Pugh Class A.
* Barcelona Clinic Liver Cancer stage C patients with no prior systemic anticancer therapy for hepatocellular carcinoma.
* Patients with an Eastern Cooperative Oncology Group performance score of 0-1.
* Adequate Hematologic and Liver Function:

A. Hemoglobin: ≥ 9.0 g/dL B. Absolute Neutrophil Count : ≥ 1,000/mm³ C. Platelet Count: ≥ 70,000/μL D. Prothrombin Time: ≥ 70% (or Prothrombin Time INR ≤ 1.2)

* Patients with upper gastrointestinal endoscopy performed within six months prior to the start of anticancer treatment.
* No plans for breastfeeding, and if of childbearing potential, using contraception or no plans for spouse's pregnancy or practicing contraception.
* Patients who have received an explanation of the treatment purpose and methods and have provided informed consent for the treatment.

Exclusion Criteria:

* Participants who have previously received systemic anticancer therapy for advanced hepatocellular carcinoma.
* Patients with intrahepatic tumor involvement of 50% or more.
* Patients with tumor thrombus in the main portal vein or both first-order branches (Vp4).
* Patients with a prior history of liver transplantation.
* with uncontrolled malignant tumors other than HCC at the time of enrollment (participation is allowed if disease-free survival exceeds two years).
* Patients with uncontrolled or serious underlying diseases requiring treatment.
* Patients with a history of esophageal or gastric variceal bleeding.
* Previous Variceal Treatments: Patients who have undergone any of the following treatments for variceal bleeding:

A. Endoscopic Variceal Obliteration (EVO) B. EVL C. Transjugular Intrahepatic Portosystemic Shunt (TIPS) D. Percutaneous Approach for Retrograde Transvenous Obliteration (PARTO) E. Surgical procedures

* Patients who have used anticoagulants or antiplatelet agents within one week prior to the study.
* Presence of grade 2 or higher isolated gastric varices or Red Color Signs confirmed by baseline endoscopy (EGD).
* Patients who are pregnant.
* Patients who are unable to understand or provide written informed consent.
* Patients deemed unsuitable for clinical study participation based on the investigator's judgment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of esophageal variceal bleeding at 6 months | From the first Atezo/Bev treatment date until the date of first esophageal varix bleeding, Atezo/Bev treatment discontinuation, or last follow-up, whichever came first, assessed up to 6 months
  The incidence of esophageal variceal bleeding at 6 months following treatment in patients with HCC receiving atezolizumab and bevacizumab as standard therapy.

SECONDARY OUTCOMES:
Cumulative incidence of acute esophageal varix bleeding | from the date of the first Atezo/Bev treatment date until the date of first esophageal varix bleeding, the discontinuation of Atezo/Bev treatment or last follow-up, whichever came first, assessed up to 12 months
  Cumulative incidence of acute esophageal varix bleeding after initiation of Atezo/Bev: acute esophageal varix bleeding is defined as:
  i) Current oozing or spurting type bleeding on the esophageal varix ii) Stigmata suggesting recent bleeding (pin-point ulceration on the varix, adherent clot, or white protrusion in the setting of hematemesis but no other cause of UGI bleeding) iii) Post-EVL ulcer bleeding is also considered esophageal varix bleeding
Cumulative incidence of non-variceal GI bleeding | from the date of the first Atezo/Bev treatment date until the date of first non-variceal GI bleeding, the discontinuation of Atezo/Bev treatment or last follow-up, whichever came first, assessed up to 12 months
  non-variceal GI bleeding is defined as new-onset hematemesis, melena or both combined with overall hemorrhage from the upper GI tract except for esophageal varix bleeding
Overall survival | from the date of the first Atezo/Bev treatment date until the date of death, the discontinuation of Atezo/Bev treatment or last follow-up, whichever came first, assessed up to 12 months
  Overall survival will be evaluated
Cumulative incidence of liver-related complications (except for esophageal varix bleeding) | from the date of the first Atezo/Bev treatment date until the date of first liver-related complications (except for esophageal varix bleeding), the discontinuation of Atezo/Bev treatment or last follow-up, whichever came first, assessed up to 12 months
  liver-related complication is defined as ascites, spontaneous bacterial peritonitis, and hepatic encephalopathy
Incidence of EVL-related complications | from the date of the first Atezo/Bev treatment date until the date of first EVL-related complications, the discontinuation of Atezo/Bev treatment or last follow-up, whichever came first, assessed up to 12 months
  EVL-related complications will be evaluate after initiation of first EVL
Quality of Life Assessment Related to Treatment | Before the date of first EVL, first Atezo/Bev treatment date, and first/third EGD surveillance after first EVL
  Patient-reported outcomes will be assessed using validated QoL instruments that are widely used in clinical trials for HCC and systemic therapy:
  1. EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) Scoring: Each domain is scored on a 0-100 scale, with higher scores in functional scales indicating better QoL, while higher scores in symptom scales indicate greater symptom burden.
  2. EORTC QLQ-HCC18 (HCC-Specific Module) Scoring: Symptoms are rated on a scale of 1 to 4 (1 = not at all, 4 = very much). Higher scores indicate worse symptoms.
Development of biomarker predicting occurrence of variceal bleeding and clinical outcome | through 24 weeks
  A total of 20 mL of peripheral blood will be collected. If these samples are not collected during the scheduled visits, they may be obtained at any time during the clinical trial. Additional samples may also be collected depending on the patient's clinical condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jihyun An, MD, PhD, Study Director — Gastroenterology and Hepatology, Hanyang University College of Medicine, Guri, Republic of Korea
Locations (1):
- Liver cancer center, Asan Medical Center, Seoul, Song-pa, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Singal AG, Llovet JM, Yarchoan M, Mehta N, Heimbach JK, Dawson LA, Jou JH, Kulik LM, Agopian VG, Marrero JA, Mendiratta-Lala M, Brown DB, Rilling WS, Goyal L, Wei AC, Taddei TH. AASLD Practice Guidance on prevention, diagnosis, and treatment of hepatocellular carcinoma. Hepatology. 2023 Dec 1;78(6):1922-1965. doi: 10.1097/HEP.0000000000000466. Epub 2023 May 22. No abstract available. PMID 37199193
- [Result] Ben Khaled N, Moller M, Jochheim LS, Leyh C, Ehmer U, Bottcher K, Pinter M, Balcar L, Scheiner B, Weich A, Leicht HB, Zarka V, Ye L, Schneider J, Piseddu I, Ocal O, Rau M, Sinner F, Venerito M, Gairing SJ, Forster F, Mayerle J, De Toni EN, Geier A, Reiter FP. Atezolizumab/bevacizumab or lenvatinib in hepatocellular carcinoma: Multicenter real-world study with focus on bleeding and thromboembolic events. JHEP Rep. 2024 Apr 8;6(6):101065. doi: 10.1016/j.jhepr.2024.101065. eCollection 2024 Jun. PMID 38798717
- [Result] Ha Y, Kim JH, Cheon J, Jeon GS, Kim C, Chon HJ. Risk of Variceal Bleeding in Patients With Advanced Hepatocellular Carcinoma Receiving Atezolizumab/Bevacizumab. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2421-2423.e2. doi: 10.1016/j.cgh.2022.07.035. Epub 2022 Aug 6. No abstract available. PMID 35944830
- [Result] Song YG, Yeom KM, Jung EA, Kim SG, Kim YS, Yoo JJ. Risk of Bleeding in Hepatocellular Carcinoma Patients Treated with Atezolizumab/Bevacizumab: A Systematic Review and Meta-Analysis. Liver Cancer. 2024 May 22;13(6):590-600. doi: 10.1159/000539423. eCollection 2024 Dec. PMID 39687040
- [Result] Jaiswal V, Jain E, Hitawala G, Loh H, Patel S, Thada P, Nandwana V, Pandey S, Quinonez J, Naz S, Stein JD, Cueva W. Bevacizumab and Sinus Venous Thrombosis: A Literature Review. Cureus. 2021 Nov 11;13(11):e19471. doi: 10.7759/cureus.19471. eCollection 2021 Nov. PMID 34912612
- [Result] Patel JN, Jiang C, Owzar K, Hertz DL, Wang J, Mulkey FA, Kelly WK, Halabi S, Furukawa Y, Lassiter C, Dorsey SG, Friedman PN, Small EJ, Carducci MA, Kelley MJ, Nakamura Y, Kubo M, Ratain MJ, Morris MJ, McLeod HL. Pharmacogenetic and clinical risk factors for bevacizumab-related gastrointestinal hemorrhage in prostate cancer patients treated on CALGB 90401 (Alliance). Pharmacogenomics J. 2024 Mar 4;24(2):6. doi: 10.1038/s41397-024-00328-z. PMID 38438359
- [Result] Cheng AL, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Lim HY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Ma N, Nicholas A, Wang Y, Li L, Zhu AX, Finn RS. Updated efficacy and safety data from IMbrave150: Atezolizumab plus bevacizumab vs. sorafenib for unresectable hepatocellular carcinoma. J Hepatol. 2022 Apr;76(4):862-873. doi: 10.1016/j.jhep.2021.11.030. Epub 2021 Dec 11. PMID 34902530
- [Result] Larrey E, Campion B, Evain M, Sultanik P, Blaise L, Giudicelli H, Wagner M, Cluzel P, Rudler M, Ganne-Carrie N, Thabut D, Allaire M. A history of variceal bleeding is associated with further bleeding under atezolizumab-bevacizumab in patients with HCC. Liver Int. 2022 Dec;42(12):2843-2854. doi: 10.1111/liv.15458. Epub 2022 Oct 26. PMID 36254617

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT06819566/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT06819566/ICF_001.pdf